CLINICAL TRIAL: NCT00609154
Title: Effect of GLP-1 on Insulin Biosynthesis and Turnover Rates
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per source documents the study was terminated well in advance of targeted enrollment. A method for the analysis of insulin and proinsulin samples was never fully developed and validated. Study terminated upon expiration of IRB approval
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1999-041, Sub-study #4; Sub-study 4 (Other: Merck Sharp & Dohme Corp.); R01DK061644-09 (NIH)
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Insulin; biosynthesis; Non diabetic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Glucagon-Like Peptide 1; Incretins; Glycemic Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetic Group (Experimental): Participants with Type 2 diabetes
  Interventions: Drug: glucagon like peptide-1; Dietary Supplement: glucose control
- Non-diabetic Group (Active Comparator): Participants who are non-diabetic will serve as control. treatment is matched to experimental group
  Interventions: Drug: glucagon like peptide-1; Dietary Supplement: glucose control

INTERVENTIONS:
Drug: glucagon like peptide-1 — GLP-1 1 pmole/kg/min
  Other Names: incretin
Dietary Supplement: glucose control — glucose without GLP-1

SUMMARY:
The gut hormone glucagon like peptide-1 (GLP-1) has been shown to have important effects on maintaining the function and health of the insulin producing beta cells. This hormone is known to increase the production rate of new insulin as well as increase the release of insulin into the blood.

DETAILED DESCRIPTION:
We will measure the rate of new insulin production in subjects with Type 2 diabetes compared to non diabetic subjects. We hypothesize that subjects with Type 2 diabetes make less insulin in response to GLP-1 compared to non diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Non diabetic

Exclusion Criteria:

* Currently taking medication such as thiazolidinediones, metformin, Exenatide, or sitagliptin
* Chronic condition such as chronic heart failure CHF), Coronary Artery Disease (CAD), or chronic renal failure (CRF)
* Anemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08-12 (Actual); Primary Completion 2014-05-13 (Actual); Study Completion 2014-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Stein, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicinie, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of study participants across the range of 1999-041 studies occurred at the Albert Einstein College of Medicine beginning in November 2007. The first participant into 1999-041, Substudy #4 was enrolled during August 2010.
Pre-assignment Details: Of the 22 participants who provided informed consent for 1999-041 Substudy #4, 20 met inclusion/exclusion criteria and were enrolled and randomized into the study.
Period: Overall Study
Arm/Group | Diabetic Group | Non-diabetic Group
Started | 3 | 17
Completed | 2 | 9
Not Completed | 1 | 8
Not completed — Protocol Violation | 1 | 2
Not completed — Unable to establish IV access | 0 | 4
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetic Group | Non-diabetic Group | Total
Number analyzed (Participants) | 3 | 17 | 20
Age, Customized [Count of Participants; unit: Participants]
  20-29 years old | 0 | 3 | 3
  30-39 years old | 0 | 5 | 5
  40-49 years old | 3 | 5 | 8
  50-59 years old | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 1 | 10 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 7 | 9
  Hispanic or Latino | 1 | 4 | 5
  White, Not Hispanic | 0 | 4 | 4
  Asian | 0 | 0 | 0
  Multiracial | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 17 | 20

OUTCOME MEASURES:

1. Primary Outcome: Insulin Biosynthesis Rate
Description: Blood insulin biosynthesis rate
Time Frame: 24 hours
Population: Study was terminated early. The LC/MS assay being developed to optimize and validate the analysis of insulin and proinsulin biosynthesis samples was never completed and, as such, data were not collected.
Arm/Group | Diabetic Group | Non-diabetic Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were evaluated for adverse events during the course of each IV infusion date. Infusion dates took placed during study visits and were up to 4 full days in duration, scheduled up to 1 year based on availability
Arm/Group | Diabetic Group | Non-diabetic Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/17
Other Adverse Events (participants affected / at risk) | 0/3 | 7/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetic Group (N=3) | Non-diabetic Group (N=17)
Muscle Cramp (transient) (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 — Thighs/toes
Superficial Thrombophlebitis (Vascular disorders) | 0 | 1 — Nodules
Nausea (Gastrointestinal disorders) | 0 | 5
Vomiting (Gastrointestinal disorders) | 0 | 4
Fever (General disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 — Unconfirmed
Bruising (Injury, poisoning and procedural complications) | 0 | 1 — Ecchymosis
Edema Limbs (General disorders) | 0 | 1 — Left arm swelling
Injection Site Reaction (General disorders) | 0 | 1 — Blistering adjacent to IV site
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No